CLINICAL TRIAL: NCT03104244
Title: Longitudinal Brain Health in Youth Tackle Football Players
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: More Foundation (Other)
Collaborators: Riddell, LLC (Unknown); ElMindA Ltd (Industry); Mimic Systems (Other)
Responsible Party: Principal Investigator, Sean Rose, M. D., Director of Clinical Research and Regional Director, The CORE Institute
Other Study IDs: MoreFoundation
Record Dates: First submitted 2016-09-12; First posted 2017-04-07 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Concussion, Brain; Athletic Injuries
Keywords: concussion; subconcussive impacts; brain function; football
MeSH Terms: conditions — Brain Concussion; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Youth Football: 5th and 6th grade tackle football players will be enrolled in 2016. They will be followed as a cohort, participating in the study each year they play tackle football, through 8th grade. Total enrollment is expected to reach 70 players.
- High School Football: Varsity football players from Brighton High School are eligible for the study in each year of the study. The varsity team consists of approximately 80 players. Total enrollment in this group is expected to reach 200 subjects; 80 the first year with 40 additional enrolled each subsequent year of the study.

SUMMARY:
The purpose of this study is to determine the neurologic and cognitive effects of playing tackle football in grade school and high school.

During contact practices and games, players wear a football helmet containing an impact sensor. Before and after each season, players complete neurological testing to measure several different aspects of brain function.

Two groups of football players will be in the study:

5th and 6th grade tackle football players from the Brighton Bulldogs Football and Cheer league (about 70 players).

Varsity football players from Brighton High School (about 70 players per year).

The study begins in July 2016 and will continue for 4 years (through the winter of 2020).

DETAILED DESCRIPTION:
Football players wear a football helmet containing the InSite Impact Response System that measures when, how hard, and where the helmet is hit. Coaches (or athletic trainer) are notified of threshold impacts via a sideline handheld device.

Each year pre and post-season, subjects will complete several tests of brain function during a clinic visit. These tests are listed in the "secondary outcomes" section.

Specific Aims:

1. To quantify the cumulative head impact burden during consecutive seasons of youth tackle football and high school football.
2. To detect impairment in neurologic and cognitive function from playing youth tackle football and high school football.
3. To use cumulative head impact burden to predict the development of neurologic and neurocognitive impairment.
4. To compare the effect of head impacts on youth tackle football players verses high school football players.

ELIGIBILITY:
Inclusion Criteria:

* Male football players 9-19 years of age at time of enrollment.
* Youth Football:
* 5th and 6th grade tackle football players from the Brighton Bulldogs Football and Cheer league.
* High School Football:
* Varsity Brighton High School football players.

Exclusion Criteria:

* History of moderate or severe traumatic brain injury. This is defined as loss of consciousness >30 minutes or amnesia >24 hours.
* Hearing problem preventing completion of the study testing.
* Legal blindness, preventing completion of the study testing.
* Non-English speaking subjects, preventing completion of the study testing.
* Ward of the State.

Ages: 9 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth and high school football players from teams included in the study
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Impact Monitoring (g force) | The football season runs from early August through late October or November (3-4 months)
  Each subject in the study group will be fitted with a football helmet containing the InSite impact response system. Subjects will be monitored for impacts during all contact practices and games.

SECONDARY OUTCOMES:
Neurological history | Occurs pre-season & post season and continues for 4 years
  Determine family and personal neurological history of the subject
Neurological physical examination | Occurs pre-season & post season and continues for 4 years
  Physician performed neurological examination
Cogstate | Occurs pre-season & post-season and continues for 4 years
  Brief computerized neurocognitive test
Pen and paper neuropsychological tests | Occurs pre-season & post-season and continues for 4 years
  Pen and paper tasks that assess memory, attention, and processing
Brain Network Activation (BNA) EEG test | Occurs pre-season & post-season and continues for 4 years
  evoked-response electroencephalogram
Vestibular/Ocular Motor Screening (VOMS) test | Occurs pre-season & post-season and continues for 4 years
  Assessment of eye movements and associated symptoms of headache, dizziness, nausea, and fogginess
MimicBalance! | Occurs pre-season & post-season and continues for 4 years
  video capture balance test that incorporates several different postures, including BESS postures
Strength and Difficulties Questionnaire | Occurs pre-season & post-season and continues for 4 years
  Self assessment questionnaire
SWAN ADHD Questionnaire | Occurs pre-season & post season and continues for 4 years
  Strengths and weaknesses of ADHD symptoms and normal behavior (SWAN) questionnaire completed by parent or legal guardian.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Rose, M.D., Principal Investigator — The Sports Neurology Clinic
Locations (1):
- The Sports Neurology Clinic at the CORE Institute, Brighton, Michigan, United States

IPD SHARING:
Plan to Share IPD: No